CLINICAL TRIAL: NCT04040023
Title: Optimization of Transfusion Use and Interest of the Correction of Iron Deficiencies in Cardiac Surgery Under Extracorporeal Circulation (ECC)
Brief Title: Patient Blood Management in Cardiac Surgery
Acronym: PBMc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Dr Hélène Charbonneau, Principal investigator, MD, PhD, Clinique Pasteur
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2019-A01522-55
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Surgical Blood Loss
Keywords: Red Blood Cell transfusion; Anemia; Iron deficiency; Extracorporeal circulation or Bypass; Cardiac Surgery
MeSH Terms: conditions — Blood Loss, Surgical; Anemia; Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Intervention Model Description: Prospective monocentric superiority study in two successive steps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I Group: PBMi (Other): Non-drug intervention First part of PBM program (PBMi) Training part for medical care staff to improve transfusion practices
  Interventions: Other: PBMi: Training program to improve transfusion practices
- C Group: PBMc (Experimental): Patient Blood Management: full program
  PBMi intervention and Drug intervention (systematic correction of pre- and postoperative iron and vitamin deficiencies, and erythropoietin preoperative treatment for anemic patient)
  Interventions: Drug: Iron and vitamin Deficiencies Correction Program; Other: PBMi: Training program to improve transfusion practices

INTERVENTIONS:
Drug: Iron and vitamin Deficiencies Correction Program — Preoperative:
  For patient with iron deficiency: Intravenous iron supplementation For patient with folic acid or vitamin B12 deficiency : oral vitamin supplementation For patient with anemia: pre operative erythropoietin injections
  Postoperative:
  Systematic iron supplementation
  Arms: C Group: PBMc
Other: PBMi: Training program to improve transfusion practices — Training program to sensitize health care staff to streamline the use of transfusion targeting the following points: limit perioperative and post operative hemodilution; to adapt the transfusion threshold to the tolerance of the patient to anemia in per and postoperative; justify the use of RBC transfusion by setting up a questionnaire; encourage transfusion of RBC unit by unit.

SUMMARY:
Preoperative anemia is associated with an important increase in transfusions of red blood cells (RBC) compared to a non-anemic patient in cardiac and non cardiac surgery. Furthermore transfusion is also an independent factor of morbi-mortality with notably an increase in the infectious risk, immunological, an increase of the risk of cardiac decompensation, respiratory decompensation Transfusion Related Acute Lung Injury (TRALI) or Transfusion Associated Cardiac Overload (TACO), and an increase in mortality of 16%.

Management of perioperative transfusion is therefore a public health issue. Since 2010, the World Health Organization (WHO) has been promoting a systematic approach to implement blood management programs for the patient to optimize the use of resources and promote quality and safety of care.

Improving the relevance of transfusion in cardiac surgery could be achieved by optimizing the management of patients around 2 axis:

A:non-drug intervention : Review of Practices to Improve the Management of Perioperative RBC Transfusion

B:drug intervention : Systematic correction of pre- and postoperative iron, vitamin deficiencies and anemia

The aim of this program is to improve the relevance of transfusion in cardiac surgery and to limit the morbidity and mortality induced by transfusion. This program is part of a global project of pre, per and postoperative management of the patient undergoing cardiac surgery programmed under extracorporeal circulation (ECC). It requires a multidisciplinary approach between cardiologists, anesthesiologists and intensivists, perfusionists, cardiac surgeons and paramedical teams to optimize the management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for cardiac surgery under ECC
* Patient affiliated or beneficiary of a social security scheme
* Patient having given his consent

Exclusion Criteria:

* Urgent surgery (less than 48h)
* Contraindication to iron injection : proven allergic reaction
* Erythropoietin allergy
* Protected patients: Majors under some form of guardianship or other legal protection; pregnant, breastfeeding or parturient woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
RBC transfusion rate | Between surgery and hospital discharge, an average of 10 days
  Proportion of patient who received at least one RBC transfusion during their hospitalization

SECONDARY OUTCOMES:
Adverse events | between baseline (1 month before surgery) and 3 months after surgery
  Occurrence of adverse event
Transfusion parameters | between surgery and hospital discharge, an average of 10 days
  Transfusion rate, use of poly transfusion, hemodilution, transfusion thresholds and postoperative bleeding volume.
Blood test parameters | between baseline (1 month before surgery) and 3 months after surgery
  hemoglobin, ferritin
6 min walk test | at discharge of the healthcare and rehabilitation units
  Walking test : distance reach after 6 min
New York Heart Association (NYHA) | between baseline (1 month before surgery) and 3 months after surgery
  NYHA Functional Classification
Euro Quality of life 5 dimensions (EQ5D) | between baseline (1 month before surgery) and 3 months after surgery
  EQ5D Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Charbonneau, MD, PhD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

REFERENCES:
- [Derived] Charbonneau H, Pasquie M, Savy N, Mayeur N. Hemoglobin Optimization and Transfusion Reduction Through Anemia and Iron Deficiency Correction: A Post Hoc Prospective Study in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2025 Nov 24:S1053-0770(25)01164-4. doi: 10.1053/j.jvca.2025.11.028. Online ahead of print. PMID 41483954
- [Derived] Charbonneau H, Pasquie M, Berthoumieu P, Savy N, Autones G, Angles O, Berthelot AL, Croute-Bayle M, Decramer I, Duterque D, Gabiache Y, Julien V, Mallet L, M'rini M, Quedreux JF, Richard B, Sidobre L, Taillefer L, Soula P, Garcia O, Abouliatim I, Vahdat O, Bousquet M, Ferradou JM, Jansou Y, Brunel P, Breil C, Mayeur N. Patient blood management in elective bypass cardiac surgery: A 2-step single-centre interventional trial to analyse the impact of an educational programme and erythropoiesis stimulation on red blood cell transfusion. Contemp Clin Trials Commun. 2020 Jul 15;19:100617. doi: 10.1016/j.conctc.2020.100617. eCollection 2020 Sep. PMID 32695923